CLINICAL TRIAL: NCT04787588
Title: COVID-19 Infection and Epithelial Cell Markers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Gail Gauvreau, Professor Department of MEdicine, McMaster University
Other Study IDs: 11033-T
Record Dates: First submitted 2021-03-04; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Asthma; Covid19
MeSH Terms: conditions — Asthma; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood TSLP levels will be measured and SNP genotyping for alarmins will be performed from Cohort 1 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospitalized patients: 100 patients hospitalized with Covid-19, and 100 hospitalized controls without Covid-19
- Mild/Moderate asthma and health controls: 20 asthmatic patients, 10 patients with asthma and allergic rhinitis, and 5 healthy controls.

SUMMARY:
To assess if TSLP expression by airway epithelial cells following COVID-19 infection regulates viral load and disease severity.

DETAILED DESCRIPTION:
The study aim is to determine the relationship between COVID-19 infection and epithelial cell expression of TSLP. Two cohorts will be used. Cohort One will include 100 hospitalized patients with Covid-19, and 100 hospitalized patients without Covid-19. Cohort 2 will include mild/moderate asthmatics and healthy controls with bio-banked biopsy material used from donors who have previously consented for samples to be used for future research.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above;
* Able to give informed consent;
* Clinically tested for SARS-CoV-2 (as completed by standard laboratory testing e.g. RT-PCR) and with a positive result and clinical features in keeping with COVID-19 illness. The control group will be patients with a negative RT-PCR COVID-19 test and without any clinical features to suggest COVID-19 illness. In addition, the control group should have NO known or current features of respiratory infection, COPD, asthma, interstitial lung disease, other respiratory inflammatory conditions or lung cancer.
* Able to provide a breath sample (as based on clinical judgement).

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 235 (Estimated)
Dates: Start 2021-02-14 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
TSLP expression in nasal epithelium | Through study completion, an average of 1 year
  Compare the level of TSLP expression in nasal epithelium in patients with and without COVID-19 infection

SECONDARY OUTCOMES:
TSLP expression in endobronchial biopsies | Baseline
  Epithelial cell expression (protein staining) of TSLP in endobronchial biopsy tissue of asthmatic patients versus normal controls.
IL-33 expression in endobronchial biopsies | Baseline
  Epithelial cell expression (protein staining) of IL-33 in endobronchial biopsy tissue of asthmatic patients versus normal controls.
ACE-2 receptor expression in endobronchial biopsies | Baseline
  Epithelial cell expression (protein staining) of ACE-2 receptor in endobronchial biopsy tissue of asthmatic patients versus normal controls.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Gauvreau, PhD, Principal Investigator — McMaster University Hospital
Locations (1):
- McMaster Cardio-Respiratory Research Lab, Hamilton, Ontario, Canada